CLINICAL TRIAL: NCT05982314
Title: A Safety and Immunogenicity Extension Study of GPNV-001
Brief Title: Extension Safety and Immunogenicity Study of GPNV-001
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GPN Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GPNV-002
Record Dates: First submitted 2023-07-24; First posted 2023-08-08 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Gamma-PN3 50 mcg (Experimental): In GPNV-001 participants will have received 2 doses of 50 mcg Gamma-PN3 at intervals of 4 weeks
  Interventions: Biological: Gamma-PN3
- Gamma-PN3 250 mcg (Experimental): In GPNV-001 participants will have received 2 doses of 250 mcg Gamma-PN3 at intervals of 4 weeks
  Interventions: Biological: Gamma-PN3
- Gamma-PN3 1000 mcg (Experimental): In GPNV-001 participants will have received 2 doses of 1000 mcg Gamma-PN3 at intervals of 4 weeks
  Interventions: Biological: Gamma-PN3
- Pneumovax 23 (Active Comparator): In GPNV-001 participants will have received one 0.5ml dose of Pneumovax-23 followed by saline placebo 4 weeks later
  Interventions: Biological: Pneumovax-23
- Prevenar-13 (Active Comparator): In GPNV-001 participants will have received one 0.5ml dose of Prevenar-13 followed by saline placebo 4 weeks later
  Interventions: Biological: Prevenar-13
- Placebo (Placebo Comparator): In GPNV-001 participants will have received two doses of 0.5 ml saline placebo at intervals of 4 weeks.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Gamma-PN3 — Experimental whole-cell pneumococcal vaccine
  Arms: Gamma-PN3 1000 mcg; Gamma-PN3 250 mcg; Gamma-PN3 50 mcg
Biological: Pneumovax-23 — Licensed pneumococcal vaccine
  Arms: Pneumovax 23
Biological: Prevenar-13 — Licensed pneumococcal vaccine
  Arms: Prevenar-13
Biological: Placebo — Saline placebo
  Arms: Placebo

SUMMARY:
A 6 and 12 month safety and immunogenicity study of participants in study GPNV-001, a novel whole-cell pneumococcal vaccine.

DETAILED DESCRIPTION:
A 6 and 12 month safety and immunogenicity study of participants in study GPNV-001, a novel whole-cell pneumococcal vaccine. Up to 20 participants per cohort will be invited.

ELIGIBILITY:
Inclusion Criteria:

1. Completion of study GPNV-001 as per protocol with no significant deviations.
2. Has provided written informed consent.

Exclusion Criteria:

1. Potential participants will be excluded if they have received a pneumococcal vaccine since the end of study visit for study GPNV-001
2. A potential participant has had an episode of pneumonia since completing Study GPNV-001

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Serum IgG titre to Gamma-PN3 | 6 months and 12 months
  Serum IgG titre to the vaccine
Serious adverse events | 6 months and 12 months
  Serious adverse events occurring after day 57 of study GPNV-001

SECONDARY OUTCOMES:
Opsonophagocytic antibodies to pneumococcal strains | 6 months and 12 months
  Serum OPA titres to up to 24 pneumococcal serotypes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Adelaide, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No
No plan as yet